CLINICAL TRIAL: NCT06205706
Title: Phase 1/2a Open-Label, Dose-Escalation, Multicenter, First-in-Human, Consecutive-Cohort, Clinical Trial of BI-1910, a Monoclonal Antibody to Tumor Necrosis Factor Receptor 2 (TNFR2), as a Single Agent and in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: BI-1910 as a Single Agent and in Combination With Pembrolizumab for the Treatment of Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-BI-1910-01; U1111-1293-2634 (Other: World Health Organization); 2022-503066-74-00 (Other: European Medicines Agency); KEYNOTE F82 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-12-18; First posted 2024-01-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors; Non Small Cell Lung Cancer; Hepatocellular Carcinoma
Keywords: solid tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a Phase 1/2a, open-label, dose-escalation, multicenter, FIH, consecutive-cohort, clinical trial of BI-1910, as a single agent and in combination with pembrolizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I, Part A - Dose escalation and safety of BI-1910 as single agent (Experimental): Dose escalation of BI-1910 administered as a single agent.
  Interventions: Drug: BI-1910
- Phase I, Part B - Dose escalation and safety of BI-1910 in combination with pembrolizumab (Experimental): Dose escalation of BI-1910 in combination with pembrolizumab.
  Interventions: Drug: BI-1910; Drug: Pembrolizumab
- Phase 2a, Part A - Dose expansion of BI-1910 as single agent (Experimental): BI-1910 administered as a single agent at the hypothesized recommended phase 2 dose determined in Phase 1.
  Interventions: Drug: BI-1910
- Phase 2a, Part B - Dose expansion of BI-1910 (Experimental): BI-1910 administered in combination with pembrolizumab at the respective hypothesized recommended phase 2 doses determined in Phase 1
  Interventions: Drug: BI-1910; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BI-1910 — BI-1910 administered as a flat-dose IV infusion once every 3 weeks
Drug: Pembrolizumab — Pembrolizumab be administered as an IV infusion at its standard flat dose (200 mg) once every 3 weeks prior to the BI-1910 infusion
  Arms: Phase 2a, Part B - Dose expansion of BI-1910; Phase I, Part B - Dose escalation and safety of BI-1910 in combination with pembrolizumab

SUMMARY:
The goal of this first in human clinical trial is to test BI-1910 administered as single agent and in combination with pembrolizumab in subjects with advanced/metastatic solid tumors whose disease has progressed after standard therapy.

The main questions it aims to answer are:

* how safe and tolerable is BI-1910
* what is maximum tolerated or administrated dose
* to determine recommended dose for further clinical trials

Participants will receive infusions of BI-1910 alone or combination with pembrolizumab every 3 weeks.

DETAILED DESCRIPTION:
This is a Phase 1/2a, open-label, dose-escalation, multicenter, FIH, consecutive-cohort, clinical trial of BI-1910, as a single agent and in combination with pembrolizumab, in subjects with advanced/metastatic solid tumors whose disease has progressed after standard therapy.

The trial comprises 2 phases: a Phase 1 with Parts A and B, and a Phase 2a with Parts A and B.

Phase 1 Part A consists of a dose escalation of BI-1910 as a single agent to evaluate safety and tolerability and to determine the RP2D as a single agent (sRP2D) in subjects with advanced/metastatic solid tumors whose disease has progressed after standard therapy.

Phase 1 Part B consists of a dose escalation of BI-1910 in combination with pembrolizumab to evaluate the safety and tolerability of the combination treatment and to allow selection of the RP2D for BI-1910 in combination with pembrolizumab (cRP2D) in subjects with advanced/metastatic solid tumors whose disease has progressed after standard therapy.

Phase 2a will assess BI-1910 administered as a single agent (Part A) and in combination with pembrolizumab (Part B) at the respective hypothesized RP2D(s) determined in Phase 1. Phase 2a expansion will be conducted in indication specific cohorts of subjects. The aim of the Phase 2a is to urther assess the safety and tolerability of BI-1910 as a single agent (Part A) and in combination with pembrolizumab (Part B), characterize its PK and pharmacodynamics, and assess preliminary antitumor activity by ORR, DoR, and progression-free survival (PFS), as measured by RECIST v1.1 and iRECIST.

ELIGIBILITY:
Inclusion Criteria:

1. Is willing and able to provide signed informed consent for the trial.
2. Is ≥18 years of age on the day of signing the informed consent form.
3. Has a histologically-confirmed advanced/metastatic solid tumor.
4. Has received standard of care and progressed or is intolerant of, or is not eligible to receive standard of care antineoplastic therapy.
5. Has at least 1 measurable disease lesion as defined by RECIST v1.1.
6. Must be willing to provide tumor biopsies as specified in the schedule of assessments
7. Has a life expectancy of ≥12 weeks.
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Has adequate organ function as confirmed by laboratory values.

Exclusion Criteria:

1. Needs doses of prednisolone >10 mg daily (or equipotent doses of other corticosteroids) while on the trial other than as premedication.
2. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Has known or suspected hypersensitivity to BI-1910 or pembrolizumab.
4. Has cardiac or renal amyloid light-chain amyloidosis.
5. Has received the following:

   1. Chemotherapy or small molecule anti-cancer therapy products within 4 weeks, or 5 half-lives of the respective drug whichever is longer, of first dose of BI-1910.
   2. Radiotherapy within 2 weeks of first dose of BI-1910. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) for non-CNS disease.

      Subjects who have previously had radiation pneumonitis are not allowed.
   3. Immunotherapy within 4 weeks prior to the first dose of BI-1910.
6. Has not recovered from AEs to at least Grade 1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (v5.0 or higher).
7. Has had Grade ≥3 autoimmune manifestations of previous immune checkpoint inhibitor treatments (e.g., anti-PD-1, anti-PD-L1, or anti-CTLA-4).
8. Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
9. Has an active, known, or suspected autoimmune disease.
10. Is a female subject and has the ability to become pregnant (or already pregnant or lactating/breastfeeding). However, those female subjects who have a negative serum or urine pregnancy test up to 72 hours prior to their first dose of study treatment and agree to use a highly effective method of birth control for 4 weeks before entering the trial, during the trial, and for 12 months after their last dose of study treatment are considered eligible.
11. Is a male subject with partner(s) of childbearing potential (unless he agrees to use a barrier method of contraception [condom plus spermicidal gel] with the female partner(s) who are using one highly effective method of contraception during the trial and for 12 months after completing treatment).
12. Has had major surgery from which the subject has not yet recovered.
13. Is at high medical risk because of nonmalignant systemic disease including severe active infections on treatment with antibiotics, antifungals, or antivirals other than the ones considered adequate for treatment of HBV.
14. Has presence of chronic graft versus host disease.
15. Has had an allogenic tissue/solid organ transplant.
16. Is positive for Human Immunodeficiency Virus (HIV).
17. Has history of chronic HBV or HCV infections.
18. Has a history of active tuberculosis (Bacillus tuberculosis).
19. Has received a live vaccine within 30 days before the first dose of study treatment.
20. Has uncontrolled or significant cardiovascular disease.
21. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the trial.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
23. Is participating or planning to participate in another interventional clinical trial or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study treatment.
24. Has a known additional malignancy of another type, with the exception of adequately treated cone-biopsied carcinoma in situ and basal or squamous cell carcinoma of the skin. Male subjects with asymptomatic prostate cancer without known metastatic disease and with no requirement for therapy or requiring only hormonal therapy and with normal prostate-specific antigen for >1 year prior to start of study treatment are eligible.
25. Has a confirmed diagnosis of primary immunodeficiency or an acquired condition that leads to an immunodeficiency disorder or taking any other form of immunosuppressive therapy within 7 days prior the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2027-07-14 (Estimated); Study Completion 2028-11-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | From the start of the study treatment for up to 2 years and 90 days.
  AEs will be assessed by the investigators by severity and will be graded according to the NCI CTCAE v5.0 or higher and causality between AEs and the exposure to the study treatment.
Occurrence of serious adverse events (SAEs) | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  SAEs will be assessed by the investigators by severity and will be graded according to the NCI CTCAE v5.0 or higher and causality between SAEs and the exposure to the study treatment
Frequency of AEs leading to discontinuation of study treatment | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  All adverse events leading to premature study treatment discontinuation will be analyzed descriptively utilizing corresponding MedDRA, System Organ Classes, and Preferred Terms.
Frequency of dose interruptions and dose reductions. | From the start of the study treatment for up to 2 years
  Study treatment modifications will be summarized in 2 categories: dose reduction and dose interruptions. The number and percentage of subjects who have any dose reduction or interruption and have at least 1 dose reduction or interruption will be summarized. Lastly, the primary reason for each form of study treatment modification will also be summarized.
Changes from baseline in laboratory parameters | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  These include clinical laboratory assessments (hematology, clinical chemistry, urinalysis), additional CRP assessment, coagulation, thyroid, pregnancy, and viral serology assessments Safety laboratory results will be graded by NCI CTCAE v5.0 (or higher). If no grading exists, values will be classified into low/normal/high based on laboratory normal ranges. Each parameter will be presented by descriptive statistics at each visit, including change from baseline.
Changes from baseline in temperature (C or F) | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  Temperature (C or F) will be measured in a seated or supine position after 5 minutes' rest and will be summarized by descriptive statistics at each visit, including change from baseline.
Changes from baseline in Respiratory Rate (Breaths/Min) | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  Respiratory rate (breaths/min) will be measured in a seated or supine position after 5 minutes' rest and will be summarized by descriptive statistics at each visit, including change from baseline.
Changes from baseline in Blood Pressure (mmHg) | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  Systolic and diastolic blood pressure (mmHg) will be measured in a seated or supine position after 5 minutes' rest and will be summarized by descriptive statistics at each visit, including change from baseline.
Changes from baseline in O2 Saturation (%) | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  O2 Saturation (%) will be measured in a seated or supine position after 5 minutes' rest and will be summarized by descriptive statistics at each visit, including change from baseline.
Changes from baseline in weight | From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  Weight (kg or lb) and body surface area (m2) will be collected at Screening and on each dose day before any study treatment is administered and will be summarized by descriptive statistics at each visit, including change from baseline. Height (cm or in) will be recorded at baseline only
Occurrence of dose limiting toxicities (DLTs) | During phase 1 Part A: from the first dose of BI-1910 for 21 days. During phase 1 part B: from the first dose of BI-1910 for 42 days.
  All adverse events meeting the DLT criteria will be considered a DLT potentially related to the study treatment, regardless of Investigator/Sponsor causality assessment, excluding toxicities that are clearly related to disease progression or inter-current illness. DLTs will be considered by the safety monitoring committee for the purposes of dosing decisions.
identification of dose/dose range fulfilling favorable PK and pharmacodynamic profile, with acceptable safety | During phase 2a from screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  based on the totality of the efficacy, safety, PK, and pharmacodynamic endpoints

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of BI-1910 | From the start of the study treatment for up to 2 years and 90 days.
  Maximum concentration (Cmax), obtained directly from the observed concentration-versus-time data will be determined.
Serum concentration-time curve [AUC] of BI-1910 | From the start of the study treatment for up to 2 years and 90 days.
  Area under the serum concentration-time curve will be determined.
Terminal half-life (t½) of BI-1910 | From the start of the study treatment for up to 2 years and 90 days.
  Terminal half-life will be determined, a minimum of 3 points will be used for estimation
Recommended dose range (RDR) | During phase 1 From screening for up to 28 days, throughout treatment for up to 2 years and through follow-up for up to 90 days
  RDR is defined as the range between the minimal reproducibly active dose (MRAD), and the MTD or MAD. MRAD is the lowest dose level at which subjects experience tumor shrinkage and/or relevant PK/pharmacodynamic parameters indicate biological activity.
Incidence and titer of antidrug antibodies (ADAs). | From the start of the study treatment for up to 2 years and 90 days.
  The detection and characterization of antibodies to BI-1910 will be performed. The samples collected will also be evaluated or BI-1910 serum concentration to enable interpretation of the antibody data. Antibodies may be further characterized and/or evaluated for their ability to neutralize the activity of the study treatments.
Objective response rate (ORR). | During phase 2a from from the start of the study treatment for up to 2 years and 30 days
  Objective response rate based on the best objective response, defined as achieving confirmed CR and/or PR measured by RECIST 1.1 and iRECIST,
Duration of response (DoR). | During phase 2a from from the start of the study treatment for up to 2 years and 30 days
  Defined as the time from the first assessment of PR or CR to the follow-up first assessment of PD measured by RECIST 1.1 and iRECIST.

CONTACTS AND LOCATIONS:
Overall Officials: Andres McAllister, PhD, Study Director — BioInvent International AB
Locations (8):
- Rigshospitalet, Copenhagen, Denmark
- Universitätsklinikum Essen, Essen, Germany
- Spain (4):
  - Hospital HM Nou Delfos, Barcelona
  - HM Sanchinarro, Madrid
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital universitario Virgen del Rocio, Seville
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Solna, Stockholm